CLINICAL TRIAL: NCT02714023
Title: Water And Saline Head-to-head In The Blinded Evaluation Study Trial
Acronym: WASHITBEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1201672
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Acute Appendicitis; Abscess
MeSH Terms: conditions — Appendicitis; Abscess | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Saline (Active Comparator): Patients were randomized to receive normal saline as an irrigation solution during appendectomy.
  Interventions: Procedure: Normal Saline
- Sterile Water (Active Comparator): Patients were randomized to receive sterile water as an irrigation solution during appendectomy.
  Interventions: Procedure: Sterile Water
- No irrigation used (No Intervention): Patients who do not receive any irrigation at time of operation.

INTERVENTIONS:
Procedure: Normal Saline — Intra-operative irrigation with normal saline
  Arms: Normal Saline
Procedure: Sterile Water — Intra-operative irrigation with sterile water
  Arms: Sterile Water

SUMMARY:
Patients who are diagnosed with acute appendicitis consented and then randomized into two arms of the trial. In one arm, patients receive irrigation of the abdomen during surgery with normal saline, or salt water. In the other arm, patients receive irrigation of the abdomen during surgery with sterile water. Sometimes patients receive no irrigation if none is determined to be needed at the time of operation by the surgeon. We then followed patients after surgery for 30 days. The hypothesis of this study was that the use of sterile water as irrigation fluid during surgery in patients who have acute appendicitis will decrease the chance of a post-operative abscess or infection.

DETAILED DESCRIPTION:
All patients, aged 6 and above, who present for an emergent or interval appendectomy to any one of the participating surgeons will potentially be enrolled in the study. Prior to surgery, the patient or the patient's guardian if a minor, will be informed of the study and consent (assent of minors will be obtained) will be requested. If consent is obtained, the patient's name and medical record number will then be sent to the inpatient pharmacy. They will be randomly assigned using a master list to either water or saline arm. The pharmacy will then send the correct solution to the operating room in the form of 3 one Liter bags. This will be ordered prior to going to the operating room. Next, a laparoscopic or open appendectomy will be performed according to the current standard of care. The surgeon will also be free to convert a laparoscopic procedure to an open procedure if deemed appropriate by his or her clinical judgment. The type of irrigant used during the case, however, will be blinded to the surgeon. The surgeon will use as much irrigation solution as they deem necessary based on an intra-operative decision. This will likely not have any affect on the study, as there is no standard amount of irrigation that is needed during appendectomies, and we do not wish to change the current practices of our surgeons. Additionally, the study question of if sterile water will decrease infectious rates will not be affected either. The science of this study will remain the same whether 10 mL or 3000 mL of irrigation solution is utilized. The surgeon may use more irrigation if deemed necessary to adequately wash the abdomen and remove all particulate matter and blood clots. At the end of the case, the surgeon will record the amount of irrigant used along with surgery date, duration of symptoms, surgery start and finish time, preoperative antibiotics, height and weight. The patient will be followed in the study for 30 days after surgery. There is usually a follow up office visit one to two weeks after the procedure. A chart review after the case will capture the length of stay, post-operative antibiotic, pathology report results, and complications consisting such as prolonged ileus (>2 days), bowel obstruction, prolonged fever (> 2 days), post-operative abscess, irrigation volume, and wound infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients, age 6 and older, who present for an emergent or interval appendectomy to any one of the participating surgeons, meet the inclusion criteria for the study. Assent from all minors (under age 18) was obtained.

Exclusion Criteria:

* Pregnant patients, patients with mental handicap, Veterans, patients under 6 years old

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Post-operative deep space organ infection as defined by the Surgical Infection Society | 30 days
  Infection after surgery within the peritoneal space

SECONDARY OUTCOMES:
Temperature greater than 38.5 degree Celsius | 30 days
  Chart review for evidence of prolonged fever >38.5 for >2 days
Greater than 2 days to return of bowel function as evident by either flatus or bowel movement | 30 days
  Chart review for evidence of prolonged ileus for >2days
Length of Hospital Stay | 30 days
  Medical record will be reviewed for hospital length of stay following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Rawlings, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore CB, Smith RS, Herbertson R, Toevs C. Does use of intraoperative irrigation with open or laparoscopic appendectomy reduce post-operative intra-abdominal abscess? Am Surg. 2011 Jan;77(1):78-80. PMID 21396311
- [Background] Hughes MJ, Harrison E, Paterson-Brown S. Post-operative antibiotics after appendectomy and post-operative abscess development: a retrospective analysis. Surg Infect (Larchmt). 2013 Feb;14(1):56-61. doi: 10.1089/sur.2011.100. Epub 2013 Feb 21. PMID 23427791
- [Background] Bonanni F, Reed J 3rd, Hartzell G, Trostle D, Boorse R, Gittleman M, Cole A. Laparoscopic versus conventional appendectomy. J Am Coll Surg. 1994 Sep;179(3):273-8. PMID 8069421
- [Background] Paik PS, Towson JA, Anthone GJ, Ortega AE, Simons AJ, Beart RW Jr. Intra-abdominal abscesses following laparoscopic and open appendectomies. J Gastrointest Surg. 1997 Mar-Apr;1(2):188-92; discussion 192-3. doi: 10.1016/s1091-255x(97)80108-4. PMID 9834347
- [Background] Krisher SL, Browne A, Dibbins A, Tkacz N, Curci M. Intra-abdominal abscess after laparoscopic appendectomy for perforated appendicitis. Arch Surg. 2001 Apr;136(4):438-41. doi: 10.1001/archsurg.136.4.438. PMID 11296116
- [Background] Shuler FW, Newman CN, Angood PB, Tucker JG, Lucas GW. Nonoperative management for intra-abdominal abscesses. Am Surg. 1996 Mar;62(3):218-22. PMID 8607582
- [Background] Solomkin JS, Mazuski JE, Bradley JS, Rodvold KA, Goldstein EJ, Baron EJ, O'Neill PJ, Chow AW, Dellinger EP, Eachempati SR, Gorbach S, Hilfiker M, May AK, Nathens AB, Sawyer RG, Bartlett JG. Diagnosis and management of complicated intra-abdominal infection in adults and children: guidelines by the Surgical Infection Society and the Infectious Diseases Society of America. Surg Infect (Larchmt). 2010 Feb;11(1):79-109. doi: 10.1089/sur.2009.9930. PMID 20163262
- [Background] Ingraham AM, Cohen ME, Bilimoria KY, Pritts TA, Ko CY, Esposito TJ. Comparison of outcomes after laparoscopic versus open appendectomy for acute appendicitis at 222 ACS NSQIP hospitals. Surgery. 2010 Oct;148(4):625-35; discussion 635-7. doi: 10.1016/j.surg.2010.07.025. Epub 2010 Aug 24. PMID 20797745
- [Background] Tzovaras G, Baloyiannis I, Kouritas V, Symeonidis D, Spyridakis M, Poultsidi A, Tepetes K, Zacharoulis D. Laparoscopic versus open appendectomy in men: a prospective randomized trial. Surg Endosc. 2010 Dec;24(12):2987-92. doi: 10.1007/s00464-010-1160-5. Epub 2010 Jun 15. PMID 20552369
- [Background] Guller U, Hervey S, Purves H, Muhlbaier LH, Peterson ED, Eubanks S, Pietrobon R. Laparoscopic versus open appendectomy: outcomes comparison based on a large administrative database. Ann Surg. 2004 Jan;239(1):43-52. doi: 10.1097/01.sla.0000103071.35986.c1. PMID 14685099
- [Background] Ward NT, Ramamoorthy SL, Chang DC, Parsons JK. Laparoscopic appendectomy is safer than open appendectomy in an elderly population. JSLS. 2014 Jul-Sep;18(3):e2014.00322. doi: 10.4293/JSLS.2014.00322. PMID 25392668
- [Background] Andersen BR, Kallehave FL, Andersen HK. Antibiotics versus placebo for prevention of postoperative infection after appendicectomy. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD001439. doi: 10.1002/14651858.CD001439.pub2. PMID 16034862
- [Background] van Rossem CC, Schreinemacher MH, Treskes K, van Hogezand RM, van Geloven AA. Duration of antibiotic treatment after appendicectomy for acute complicated appendicitis. Br J Surg. 2014 May;101(6):715-9. doi: 10.1002/bjs.9481. Epub 2014 Mar 26. PMID 24668341
- [Background] Cheng Y, Zhou S, Zhou R, Lu J, Wu S, Xiong X, Ye H, Lin Y, Wu T, Cheng N. Abdominal drainage to prevent intra-peritoneal abscess after open appendectomy for complicated appendicitis. Cochrane Database Syst Rev. 2015 Feb 7;(2):CD010168. doi: 10.1002/14651858.CD010168.pub2. PMID 25914903
- [Background] Parcells JP, Mileski JP, Gnagy FT, Haragan AF, Mileski WJ. Using antimicrobial solution for irrigation in appendicitis to lower surgical site infection rates. Am J Surg. 2009 Dec;198(6):875-80. doi: 10.1016/j.amjsurg.2009.09.002. PMID 19969145
- [Background] Fernandez R, Griffiths R. Water for wound cleansing. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD003861. doi: 10.1002/14651858.CD003861.pub3. PMID 22336796
- [Result] Addiss DG, Shaffer N, Fowler BS, Tauxe RV. The epidemiology of appendicitis and appendectomy in the United States. Am J Epidemiol. 1990 Nov;132(5):910-25. doi: 10.1093/oxfordjournals.aje.a115734. PMID 2239906